CLINICAL TRIAL: NCT06226428
Title: Ciclo-Ergometría en el Paciente Con Síndrome de Distrés Respiratorio Agudo
Brief Title: Cyclo-Ergometry in the Patient With Acute Respiratory Distress Syndrome
Acronym: NPIDRA2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUGI-cu
Record Dates: First submitted 2024-01-05; First posted 2024-01-26 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-12

CONDITIONS: Coronavirus
Keywords: Corticosteroids; Mobilization; Oxygenation; Cyclo-ergonometry; Acquired muscle weakness of the critically ill patient
MeSH Terms: conditions — Coronavirus Infections | interventions — Sitting Position; Standing Position; Machine Learning; Walking

STUDY DESIGN:
Intervention Model Description: Controlled pilot clinical trial, with randomized assignment to two treatment groups, the cyclo-ergometry program group and the usual treatment group (parallel). The randomization will be carried out by blocks and will be kept in the Clinical Epidemiology Unit. When the physician has a patient available to enter the study, a call will be made to the Clinical Epidemiology Service where a randomization code and the group to which he/she has been assigned will be indicated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclo-ergonometry program group (Experimental): * Mobility activities in bed (turning, pelvic elevation and sitting), standing, transfers and walking.
  * Progressive strength training of upper and lower limbs (2 days/week), by performing isometric exercises, strengthening with multi-resistance elastic bands or multi-weight dumbbells.
  * Cycloergometry, using the MotoMed Letto 2 device, with a progressive pattern, starting with 5 minutes and lasting up to 30 minutes. It will be performed once a day, during working days (Monday to Friday) until discharge from the intensive care unit, and at a modified Borg intensity of 2-3 (Light).
  Interventions: Other: Bed cyclo-ergonometry; Other: Bed mobility activities (turning, pelvic elevation and sitting), standing, transfers and walking.; Other: Progressive upper and lower limb strength training
- Usual treatment group (Active Comparator): * Mobility activities in bed (turning, pelvic elevation and sitting), standing, transfers and walking.
  * Progressive strength training of upper and lower limbs (2 days/week), by performing isometric exercises, strengthening with multi-resistance elastic bands or multi-weight dumbbells.
  Interventions: Other: Bed mobility activities (turning, pelvic elevation and sitting), standing, transfers and walking.; Other: Progressive upper and lower limb strength training

INTERVENTIONS:
Other: Bed cyclo-ergonometry — The MotoMed Letto 2 device will be used, with a progressive pattern, starting at 5 minutes and lasting up to 30 minutes. It will be performed once a day, during weekdays (Monday to Friday) until discharge from the intensive care unit, and at a modified Borg intensity of 2-3 (Light).
  Arms: Cyclo-ergonometry program group
Other: Bed mobility activities (turning, pelvic elevation and sitting), standing, transfers and walking. — Bed mobility activities (turning, pelvic elevation and sitting), standing, transfers and walking.
Other: Progressive upper and lower limb strength training — Performing isometric exercises, strengthening with multi-resistance elastic bands or multi-weight dumbbells.

SUMMARY:
In March 2020 the World Health Organization declares the Coronavirus disease pandemic 2019. Intensive Care Units deal entirely with patients with pneumonia complicated by Acute Respiratory Distress Syndrome, requiring aggressive respiratory treatments with long periods of connection to mechanical ventilation, sedation and immobilization, contributing to the onset of acquired critical patient muscle weakness (IAPD). IUCD is a frequent complication in intensive care units, with an incidence of 11-67%¹. Of multifactorial cause, immobilization or "bed-rest", the use of corticosteroids and neuromuscular blocking agents have been described as factors directly related to this syndrome.

Several studies have shown that mobilization of the patient with acute respiratory distress syndrome, even with extracorporeal membrane oxygenation, is safe, feasible and beneficial for the patient. Bedside cyclo-ergometry has been associated with a reduction in the degree of sarcopenia, contributing to the recovery of the critically ill patient. Several studies document that bed cyclo-ergometry is safe and feasible in critically ill patients within the first week of admission to intensive care, but few clinical trials exist.

DETAILED DESCRIPTION:
In March 2020 the World Health Organization declares the Coronavirus disease pandemic 2019. Intensive Care Units deal entirely with patients with pneumonia complicated by Acute Respiratory Distress Syndrome, requiring aggressive respiratory treatments with long periods of connection to mechanical ventilation, sedation and immobilization, contributing to the onset of acquired critical patient muscle weakness (IAPD).

IUCD is a frequent complication in intensive care units, with an incidence of 11-67%¹. Of multifactorial cause, immobilization or "bed-rest", the use of corticosteroids and neuromuscular blocking agents have been described as factors directly related to this syndrome. Each additional day of bed rest is associated with a 3 to 11% decrease in the strength of both peripheral and respiratory muscles, which translates into difficulty in weaning from mechanical ventilation, longer stay in the Intensive Care Unit and in the hospital in general, as well as an increase in morbidity and mortality. Similarly, in the first 24 hours after initiation of mechanical ventilation, diaphragmatic atrophy or dysfunction occurs, predisposing to prolonged mechanical ventilation. The need for ventilatory support for more than 48 hours has been associated with greater morbidity and mortality at hospital discharge, and survivors present greater disability and deterioration in their quality of life.

Several studies have shown that mobilization of the patient with acute respiratory distress syndrome, even with extracorporeal membrane oxygenation, is safe, feasible and beneficial for the patient. Most of the programs described in the literature include patients requiring extracorporeal membrane oxygenation, mainly in the pre-transplantation situation, and to a lesser extent patients with acute respiratory distress syndrome. They are characterized by the individual and progressive performance of functional activities of lesser to greater difficulty, starting with passive exercises of joint range, active and active-resisted exercises while the patients are in decubitus, progressing in some cases to sitting at the edge of the bed and less frequently to standing.

Bedside cyclo-ergometry has been associated with a reduction in the degree of sarcopenia, contributing to the recovery of the critically ill patient. Several studies document that bed cyclo-ergometry is safe and feasible in critically ill patients within the first week of admission to intensive care, but few clinical trials exist.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Alert and cooperative (RASS agitation-sedation between -1 and +1).
* Able to give informed consent (or authorize a family member) to be randomly assigned to receive the cyclo-ergometry program or conventional physiotherapy treatment.
* With or without connection to mechanical ventilation (via orotracheal tube or tracheostomy).
* Clinically stable (cardio-vascular, respiratory, neurological).
* With an inspired oxygen fraction less than or equal to 0.6 and requiring minimal ventilatory support (positive end-expiratory pressure less than or equal to 10 cm H2O).

Exclusion Criteria:

- Patients with pre-existing neuromuscular disease, spinal cord injury, cardiorespiratory arrest, stroke, patients with contraindications for mobility, pregnant women, advanced dementia or patients with life expectancy of less than 6 months or any situation that contraindicates the performance of cycloergometry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
CLINICAL ENDPOINT Age: Years completed at the time of inclusion in the study. | Until discharge from the intensive care unit
  Continuous quantitative variable.
CLINICAL ENDPOINT Sex: Dichotomous qualitative variable | Until discharge from the intensive care unit
  . Categories: Female/Male.
CLINICAL ENDPOINT Length of stay in the Intensive Care Unit: Number of days elapsed between admission and discharge from Intensive Care. | Until discharge from the intensive care unit
  Continuous quantitative variable.
CLINICAL ENDPOINT Overall length of stay in hospital: Number of days between admission and discharge. | Until discharge from the intensive care unit
  Continuous quantitative variable.
CLINICAL ENDPOINT Mechanical ventilation time:Number of days between intubation and successful weaning (defined as 48 hours of spontaneous breathing). | Until discharge from the intensive care unit
  Continuous quantitative variable.
CLINICAL ENDPOINT Adverse events: Defined as the presence during or within 10 minutes of cyclo-ergometry of any of the following. | Until discharge from the intensive care unit
  Discrete qualitative variable.
  Loss of airway or venous/arterial lines. Increased vasoactive drug dosage: more than 5 mcg/min Increase in blood pressure: above 200 mmHg for more than 2 minutes. Drop in mean arterial blood pressure: below 60 mmHg for more than 2 minutes. Heart rate: below 50 bpm or above 140 bpm for more than 2 minutes. Drop in arterial oxygen saturation: below 88% for more than one minute requiring increasing the inspired oxygen fraction by more than 1% for more than 5 minutes.
FUNCTIONAL ENDPOINT Gait capacity: Measured by the 6-minute walk test at the time of discharge from hospital. A simple and inexpensive physical capacity test. | Until discharge from the intensive care unit
  It reflects the level of physical activity in daily activities. It consists of walking as far as possible in 6 minutes, at a brisk pace without running, over a distance of about 30 metres. The main result is the distance covered and is recorded in metres. Arterial oxygen saturation and heart rate are monitored during the test. Available evidence suggests a minimum significant difference of 30 metres (25-33 metres) for adult patients with chronic respiratory disease.
FUNCTIONAL ENDPOINT Functional capacity: Measured at discharge from the Intensive Care Unit and at hospital discharge. | Until discharge from the intensive care unit
  By performing the Short Physical Performance Battery (SPPB)³, a test consisting of 3 items: balance, gait speed and getting up and sitting in a chair 5 times. It assesses balance, gait ability and lower limb strength. The total score ranges from 0 (worst) to 12 points (best). The SSPB has been shown to be a valid instrument for detecting frailty and predicting disability, institutionalisation and mortality. A total score of less than 10 indicates frailty and a high risk of disability and falls. A 1-point change in score has clinical relevance.
FUNCTIONAL ENDPOINT Peripheral muscle strength on admission-discharge from ICU and hospital discharge. | Until discharge from the intensive care unit
  Measurement of muscle strength using the Medical Research Council manual scale and using a dynamometer on admission and discharge from Intensive Care, as well as on discharge from hospital.
FUNCTIONAL ENDPOINT ICU MOBILITY SCALE (Spanish adaptation) | Until discharge from the intensive care unit
  A valid and reliable scale that assesses the mobility of critically ill patients and helps to plan individualised activity programmes to prevent acquired muscle weakness in the critically ill patient.
FUNCTIONAL ENDPOINT Modified Borg Scale | Until discharge from the intensive care unit
  Subjective assessment of perceived dyspnoea and fatigue during the training session.

CONTACTS AND LOCATIONS:
Locations (1):
- Asociación Instituto Biogipuzkoa, Donostia / San Sebastian, Guipuzcoa, Spain